CLINICAL TRIAL: NCT03031639
Title: Khon Kaen University's Thyroidectomy Registry
Status: Completed | Type: Observational
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Patorn Piromchai, Dr, Khon Kaen University
Other Study IDs: HE591517
Record Dates: First submitted 2017-01-20; First posted 2017-01-25 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Thyroid Nodule; Thyroid Neoplasms; Thyroid Cancer
Keywords: endoscopic; thyroidectomy
MeSH Terms: conditions — Thyroid Nodule; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic: This group is the patients who underwent endoscopic approaches thyroidectomy.
  Interventions: Procedure: Endoscopic approach thyroidectomy
- Conventional: This group is the patients who underwent conventional approach thyroidectomy

INTERVENTIONS:
Procedure: Endoscopic approach thyroidectomy — Thyroid surgery using endoscopy.
  Groups: Endoscopic

SUMMARY:
The endoscopic thyroidectomy approach is gaining popularity in the surgical field. This registry tries to collect the outcomes including quality of life and complication for both endoscopic and conventional thyroidectomy methods.

ELIGIBILITY:
Inclusion Criteria:

* The patients who underwent thyroidectomy at Khon Kaen University

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients who underwent thyroidectomy at Khon Kaen University
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-01-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of QOL Score at 6 months | 6 months
  Validated quality of life score(SF-36) will be measure at baseline and 6 months

SECONDARY OUTCOMES:
Change of the symptoms score | At 2, 6, 12, and 24 weeks after surgery
  The questionnaire for pain, numbness, voice, swallowing and neck movement function will be given and the patient needs to rate from 0 to 10.
Complication rate | At 2, 6, 12, and 24 weeks after surgery
  Complications after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patorn Piromchai, MD, MSc, PhD, Principal Investigator — Khon Kaen University
Locations (1):
- Department of Otolaryngology, Khonkaen University, Muang, Khonkaen, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piromchai P, Vatanasapt P, Reechaipichitkul W, Phuttharak W, Thanaviratananich S. Is the routine pressure dressing after thyroidectomy necessary? A prospective randomized controlled study. BMC Ear Nose Throat Disord. 2008 Mar 20;8:1. doi: 10.1186/1472-6815-8-1. PMID 18366712
- [Result] Piromchai P, Wijakkanalan P, Teeramatwanich W, Kasemsiri P, Laohasiriwong S, Ratanaanekchai T. Postauricular-submental approach endoscopic thyroidectomy. Clin Otolaryngol. 2018 Apr;43(2):767-769. doi: 10.1111/coa.12791. Epub 2016 Nov 27. No abstract available. PMID 27860271